CLINICAL TRIAL: NCT02447549
Title: A Randomised Phase II Trial of Adaptive Image Guided Standard or Dose Escalated Tumour Boost Radiotherapy in the Treatment of Transitional Cell Carcinoma of the Bladder
Brief Title: Study of Tumour Focused Radiotherapy for Bladder Cancer
Acronym: RAIDER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2014/10049
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Bladder Cancer
Keywords: IMRT; IGRT; Muscle invasive; Adaptive Radiotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WBRT (Active Comparator): Standard dose whole bladder radiotherapy
  Interventions: Radiation: WBRT
- SART (Experimental): Standard dose Adaptive tumour focused radiotherapy (SART)
  Interventions: Radiation: SART
- DART (Experimental): Dose escalated Adaptive tumour boost radiotherapy (DART)
  Interventions: Radiation: DART

INTERVENTIONS:
Radiation: WBRT — One RT plan with whole bladder treated to standard dose.
  Arms: WBRT
Radiation: SART — Three plans (small, medium & large) generated with the standard dose of RT focused on the tumour, sparing the normal bladder from full dose radiation. Pretreatment cone beam CTs will be used to select the best fitting of the three plans prior to treatment.
  Arms: SART
Radiation: DART — Three plans (small, medium & large) generated with a higher dose than standard focused on the tumour and the remainder of the bladder treated to the same dose as in the SART group. Pretreatment cone beam CTs will be used to select the best fitting of the three plans prior to treatment.
  Arms: DART

SUMMARY:
Bladder cancer is the seventh most common cancer in the UK, with 10,399 new cases diagnosed in 2011. In a quarter of these cases the cancer has infiltrated the muscular wall of the bladder (muscle invasive) and is life threatening. This type of bladder cancer is usually treated either with surgical removal of the bladder, or daily radiotherapy treatment (high strength xrays which kill cells), given every day for 4 or 7 weeks. RAIDER will investigate methods which have the potential to improve how well this radiotherapy works.

RAIDER is based on a study of novel radiotherapy techniques which was conducted at a single UK NHS Trust. Bladder radiotherapy is normally delivered using a single plan throughout treatment and treats the whole bladder with the same radiotherapy dose. In adaptive radiotherapy the delivery plan is chosen from 3 possible plans. In cancer (tumour) focused radiotherapy, the highest dose of the radiotherapy is aimed at the tumour within the bladder.

In RAIDER, at least 240 participants with muscle invasive bladder cancer will be in one of 3 treatment groups:

1. standard whole bladder radiotherapy
2. standard dose tumour focused adaptive radiotherapy
3. dose escalated tumour boost adaptive radiotherapy

Participants will visit the hospital 4 weeks, 3, 6, 9, 12, 18 and 24 months after radiotherapy and annually thereafter to check whether the cancer has returned and to receive treatment for any symptoms they may be experiencing.

RAIDER aims to confirm in a multicentre setting that novel techniques allow a higher radiotherapy dose than standard to be reliably targeted at the tumour within the bladder and to check that the long term side effects of the treatment are acceptable. If this is the case, results of RAIDER will be used to develop a study to establish whether dose escalated radiotherapy is better at treating bladder cancer than standard dose.

DETAILED DESCRIPTION:
RAIDER has a two stage design. Stage 1 will establish the feasibility of delivering DART in a multi-centre setting, and stage 2 will establish the toxicity of DART. 72 patients will be recruited in stage 1, with at least an additional 168 patients in stage 2 (sufficient to recruit 57 evaluable participants to the DART group in each fractionation cohort).

Both fractionation regimens in standard use in UK are included - 32f and 20f. Participants will be permitted to receive concomitant chemotherapy. Primary endpoints will be assessed in each fractionation cohort separately with the flexibility to drop either a fractionation cohort or an experimental treatment group (on advice of Independent Data Monitoring Committee) following completion of stage 1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥16 years
* Histologically or cytologically confirmed transitional cell carcinoma (TCC) of the bladder
* Unifocal bladder TCC staged T2-T4a N0 M0*
* Fit to receive a radical course of radiotherapy
* WHO performance status 0-2
* Willing and able to comply with study procedures and follow up schedule *Tumour location must be clearly visible on imagine or recorded on a surgical bladder map

Exclusion Criteria:

* Nodal or metastatic disease
* Multifocal invasive disease
* Simultaneous TCC in upper tract or urethra
* Pregnancy
* Active malignancy within 2 years of randomisation (not including non melanomatous skin carcinoma, previous non muscle invasive bladder tumours, NCCN low risk prostate cancer (T1/T2a, Gleason 6 PSA <10), in situ carcinoma of any site)
* Bilateral hip replacements
* Any other conditions that in the Principal Investigator's opinion would be a contra-indication to radiotherapy (e.g. previous pelvic radiotherapy / inflammatory bowel disease)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants meeting predefined radiotherapy dose constraints in DART group | 4-6 weeks from randomisation
  Primary outcome of stage 1 of study, predefined radiotherapy dose constraints for bladder, bowel and rectum met for medium plan in DART group.
Proportion of patients experiencing severe late side effects following radiotherapy. | 6-18 months post radiotherapy
  Primary outcome of stage 2 of study, late CTC toxicity grade 3 or higher.

SECONDARY OUTCOMES:
Clinician reported acute toxicity | 0-6 months post radiotherapy
  CTCAE v4
Patient reported outcomes- symptomatic toxicity | 0-24 months post radiotherapy
  Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaire
Patient reported outcomes- urinary side effects | 0-24 months post radiotherapy
  King's Health Questionnaire (KHQ)
Patient reported outcomes- sexual function | 0-24 months post radiotherapy
  excerpt of the EORTC QLQ-BLM30 questionnaire
Patient reported outcomes- chronic gastrointestinal symptoms | 0-24 months post radiotherapy
  Assessment of Late Effects of RadioTherapy - Bowel (ALERT-B) questionnaire
Patient reported outcomes- health status | 0-24 months post radiotherapy
  EQ-5D questionnaire
Loco-regional MIBC control | 0-5 years post radiotherapy
  Control of existing MIBC
Progression free survival | 0-5 years post radiotherapy
  Freedom from progressive disease
Overall survival | 0-5 years post radiotherapy
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Robert Huddart, Principal Investigator — Institute of Cancer Research/RMNHSFT
Locations (49):
- Australia (7):
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Townsville General Hospital, Douglas, Queensland
  - Radiation Oncology Mater Centre QLD, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Austin Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato, Hamilton
- United Kingdom (39):
  - Torbay District General Hospital, Torquay, Devon
  - Barts Health NHS Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Nottingham University Hospital NHS Trust, Nottingham, England
  - Queen's Hospital, Barking Havering and Redbridge University Hospitals NHS Trust, Romford, Essex
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Ayr Hospital, Ayr, Scotland
  - Maidstone Hospital, Kent Oncology Centre, Adstone
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Heart of England NHS Foundation Trust, Birmingham
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Trust, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology & Oncology Centre, Brixton
  - West Suffolk Hospital, Bury St Edmunds
  - Addenbrooke's Hospital, Cambridge
  - Velindre Hospital, Cardiff and Vale NHS Trust, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - University Hospital Coventry, Coventry
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St Luke's Cancer Centre, Guildford
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Guy's and St Thomas' Hospital, London
  - Royal Marsden NHSFT, London
  - Royal Oldham Hospital, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Northern Centre for Cancer Care, Freeman Hospital,, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - The Royal Oldham Hospital, Oldham
  - Peterborough City Hospital, Peterborough
  - Queen Alexandra Hospital, Portsmouth
  - Royal Preston Hospital, Preston
  - Weston Park Hospital, Sheffield Teaching Hospitals Trust, Sheffield
  - Kings Mill Hospital, Sherwood Forest Hospitals Foundation NHS Trust, Sutton in Ashfield
  - Musgrove Park Hospital, Taunton and Somerset NHS Foundation Trust, Taunton
  - Mid Yorkshire Hospitals, Wakefield
  - Pinderfields hospital, The Mid Yorkshire Hospitals NHS Trust, Wakefield

REFERENCES:
- [Derived] Hafeez S, Warren-Oseni K, Jones K, Mohammed K, El-Ghzal A, Dearnaley D, Harris V, Khan A, Kumar P, Lalondrelle S, McDonald F, Tan M, Thomas K, Thompson A, McNair HA, Hansen VN, Huddart RA. Bladder Tumor-Focused Adaptive Radiation Therapy: Clinical Outcomes of a Phase I Dose Escalation Study. Int J Radiat Oncol Biol Phys. 2025 Jan 1;121(1):165-175. doi: 10.1016/j.ijrobp.2024.07.2317. Epub 2024 Jul 26. PMID 39069239
- [Derived] Huddart R, Hafeez S, Omar A, Alonzi R, Birtle A, Cheung KC, Choudhury A, Foroudi F, Gribble H, Henry A, Hilman S, Hindson B, Lewis R, Muthukumar D, McLaren DB, McNair H, Nikapota A, Olorunfemi A, Parikh O, Philipps L, Rimmer Y, Syndikus I, Tolentino A, Varughese M, Vassallo-Bonner C, Webster A, Griffin C, Hall E. Acute Toxicity of Hypofractionated and Conventionally Fractionated (Chemo)Radiotherapy Regimens for Bladder Cancer: An Exploratory Analysis from the RAIDER Trial. Clin Oncol (R Coll Radiol). 2023 Sep;35(9):586-597. doi: 10.1016/j.clon.2023.05.002. Epub 2023 May 9. PMID 37225552
- [Derived] Hafeez S, Lewis R, Hall E, Huddart R; RAIDER Trial Management Group. Advancing Radiotherapy for Bladder Cancer: Randomised Phase II Trial of Adaptive Image-guided Standard or Dose-escalated Tumour Boost Radiotherapy (RAIDER). Clin Oncol (R Coll Radiol). 2021 Jun;33(6):e251-e256. doi: 10.1016/j.clon.2021.02.012. Epub 2021 Mar 23. No abstract available. PMID 33766502
- [Derived] Hafeez S, Webster A, Hansen VN, McNair HA, Warren-Oseni K, Patel E, Choudhury A, Creswell J, Foroudi F, Henry A, Kron T, McLaren DB, Mitra AV, Mostafid H, Saunders D, Miles E, Griffin C, Lewis R, Hall E, Huddart R. Protocol for tumour-focused dose-escalated adaptive radiotherapy for the radical treatment of bladder cancer in a multicentre phase II randomised controlled trial (RAIDER): radiotherapy planning and delivery guidance. BMJ Open. 2020 Dec 31;10(12):e041005. doi: 10.1136/bmjopen-2020-041005. PMID 33384390
- [Derived] Hafeez S, Lewis R, Griffin C, Hall E, Huddart R. Failing to Close the Gap Between Evidence and Clinical Practice in Radical Bladder Cancer Radiotherapy. Clin Oncol (R Coll Radiol). 2021 Jan;33(1):46-49. doi: 10.1016/j.clon.2020.07.001. Epub 2020 Aug 3. No abstract available. PMID 32762980